CLINICAL TRIAL: NCT06455605
Title: Clinical Trial of D2C7-IT + 2141-V11 Combination Immunotherapy Administered Via Convection Enhanced Delivery in Non-enhancing Tumor Post-resection of Recurrent Glioblastoma, Followed by Cervical Perilymphatic Subcutaneous Injections of 2141-V11
Brief Title: D2C7-IT + 2141-V11 Combination Post-resection in rGBM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Darell Bigner (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor-Investigator, Darell Bigner, Sponsor-Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115800
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Glioblastoma IDH Wildtype
Keywords: D2C7; D2C7-IT; 2141-V11; Pro00115800; GBM; Glioblastoma; convection-enhanced delivery; CED; IDHwt
MeSH Terms: conditions — Glioblastoma | interventions — D2C7-(scdsFv)-PE38KDEL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- D2C7-IT + 2141-V11 (Experimental): Single D2C7-IT intratumoral infusion (4613.2 ng/mL in 36 mL) over 72 hours followed by an 2141-V11 infusion over 7 hours. This is followed by injections of 2141-V11 (2mg) in the cervical perilymphatic (CPLI) subcutaneous area ipsilateral to the tumor at weeks 2, 4, 7, 10 and then every 3 weeks until week 49.
  After week 49 (equivalent of 1 year of every 3 weeks CPLI of 2141-V11), patients who have completed 1 year of CPL subcutaneous injections of 2141-V11 at 2 mg every 3 weeks, who benefit from the therapy, and desire to continue on therapy, will receive CPLI of 2141-V11 at 2 mg every 4-6 weeks.
  Interventions: Drug: D2C7-IT; Drug: 2141 V11

INTERVENTIONS:
Drug: D2C7-IT — D2C7-IT will be dosed at 166,075 ng in 36 mL.
Drug: 2141 V11 — 2141-V11 will be dosed at 3 mg in 3.5 mL for CED administration. 2141-V11 in the cervical perilymphatic subcutaneous area will be dosed at 2 mg.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the combination of D2C7-IT+2141-V11 administered in the non-enhancing tumor of patients with resected recurrent glioblastoma (rGBM) via convection enhanced delivery (CED), followed by subcutaneous cervical perilymphatic injections (CPLIs) of 2141-V11 2 and 4 weeks post infusion, then every 3 weeks for a year, and every 4-6 weeks thereafter if patients benefit from therapy.

DETAILED DESCRIPTION:
Approximately 46 evaluable patients will be enrolled in this study. Enrolled patients must have previously undergone maximal safe surgical tumor resection, with histopathologic confirmation of recurrence of GBM. Post-operative MRI also must have demonstrated a residual area of non-enhancing disease (as assessed by T2/ FLAIR images) that is amenable to infusion (no larger than 3 x 3 cm of residual enhancing disease).

Study participants will receive D2C7-IT and 2141-V11 infused in the residual disease via CED followed by repeated, imaging guided injections of 2141-V11 in the cervical perilymphatic subcutaneous area ipsilateral to the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at the time of entry into the study
2. Histopathologically confirmed WHO grade 4 IDHwt GBM (high grade glioma with molecular features of glioblastoma will be eligible)
3. Karnofsky Performance Score (KPS) ≥ 70%
4. Hemoglobin ≥ 9 g/dl prior to biopsy
5. Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion.
6. Neutrophil count ≥ 1000 prior to biopsy
7. Creatinine ≤ 1.5 x normal range prior to biopsy
8. Total bilirubin ≤ 1.5 x ULN prior to biopsy (Exception: Participant has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
9. AST/ALT ≤ 2.5 x ULN
10. Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anticoagulation will be held in the perioperative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to surgical resection and biopsy.
11. Patient must have undergone resection per the recommendation of their treating physician 3-5 weeks prior to administration of D2C7-IT, and the presence of recurrent tumor must have been confirmed by histopathological analysis.
12. Able to undergo brain MRI with and without contrast

    a. Post-surgery MRI must demonstrate a residual area of non-enhancing disease that is amenable to CED infusion (no larger than 3 x 3 cm of residual enhancing disease per screening MRI)
13. Patient or partner(s) meets one of the following criteria:

    1. Non-childbearing potential (i.e. not sexually active, physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile, or any male who has had a vasectomy). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study is defined as 1 year without menses.; or
    2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g. a condom or diaphragm) used with spermicide.
14. A signed ICF approved by the IRB will be required for patient enrollment into the study. Patients must be able to read and understand the ICF and must sign the ICF indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

1. Females who are pregnant (negative pregnancy test at screening visit) or breast- feeding
2. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
3. Patients with severe, active co-morbidity, defined as follow:

   1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
   3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
   4. Patients with known lung (forced expiratory volume in the first second of expiration (FEV1) < 50%) disease or uncontrolled diabetes mellitus
   5. Patients with albumin allergy
4. Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks), or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy
5. Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy
6. Patients may not have received treatment with tumor treating fields (e.g., Optune®)

   * 1 week prior to starting the study drug
7. Patients may not be less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation
8. Patients who have not completed all standard of care treatments, including surgical procedure and radiation therapy (Please note: For patients under 65 years old, standard radiation therapy is typically at least 59 Gy in 30 fractions over 6 weeks. For patients 65 years or older, standard RT is often reduced to a minimum 40 Gy in 15 fractions over 3 weeks.)

   1. If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial
   2. If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter methylation status is unknown at time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial
9. Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of active (growing) disease (active multifocal disease); extensive subependymal disease (tumor touching subependymal space is allowed); tumor crossing the midline or leptomeningeal disease
10. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the D2C7-IT infusion
11. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
12. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
13. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months
14. Patients who cannot undergo MRI due to obesity or to having certain metal in their bodies (i.e. pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Safety | 5 years
  Describe the safety of the combination of D2C7-IT+2141-V11 administered in non-enhancing tumor of recurrent GBM patients via CED, followed by cervical perilymphatic subcutaneous injections of 2141-V11.
  The proportion of patients who experience unacceptable toxicity will be reported.
Primary Outcome - Efficacy | 6 years
  To assess overall survival defined as the time between initiation of treatment with D2C7-IT+2141-V11 and death or last follow-up if alive.
  Median overall survival will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health Clinical Trials — https://www.dukehealth.org/clinical-trials